CLINICAL TRIAL: NCT05084911
Title: A Multi-center, Randomized, Double-blind, Parallel, Placebo-Controlled, Phase III Clinical Trial to Evaluate Efficacy and Safety of Pyramax in Mild to Moderate COVID-19 Patients
Brief Title: The Efficacy and Safety of Pyramax in Mild to Moderate COVID-19 Patients (Phase3)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SP-PA-COV-301
Record Dates: First submitted 2021-10-19; First posted 2021-10-20 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
Keywords: Pyramax; Pyronaridine; Artesunate; COVID-19; Corona virus
MeSH Terms: conditions — COVID-19 | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): Pyramax tablet
  Interventions: Drug: Pyramax
- Control (Placebo Comparator): Placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyramax — Pyronaridine-Artesunate(180/60mg) tablet for 3days.
  Arms: Test
Drug: Placebo — Placebo tablet for 3days.
  Arms: Control

SUMMARY:
This study is a multi-center, randomized, double-blind, parallel, placebo-controlled, phase III clinical trial to evaluate efficacy and safety of pyramax in mild to moderate COVID-19 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females aged 19 years or older (or minimum age for adulthood or for informed consent below 19 years for each country)
2. Patients with body weight ≥45 kg at screening
3. Patients with COVID-19 confirmed by RT-PCR before randomization
4. Patients confirmed with mild or moderate COVID-19, along with one or more symptoms in association with COVID-19 within 5 days before randomization, who do not need adjunctive oxygen therapy
5. Patients who are fully informed of this study, voluntarily decide to participate in this study and provide written consent to comply with requirements for this study

Exclusion Criteria:

1. Patients with severe or critical* COVID-19
2. Patients requiring hospitalization for therapeutic purposes for COVID-19 such as oxygen therapy with a decrease of oxygen saturation (<94%) at screening or higher level of care, or who may be potentially transferred to another hospital other than the clinical trial institution within 72 hours.
3. Patients who have received or who have planned to receive any anti-viral drugs to treat COVID-19 infection or medications that may affect the course of treatment within 28 days before participating in this study or before a sufficient wash-out period [more than five times the half-life of the drug, etc.] (the longer period between the two is chosen).
4. Patients with one or more of the following infections in the past or present

   1. Infection with need for systemic anti-infection treatment other than Corona virus (SARS-CoV-2)
   2. Major infection with need for oral antibiotics or hospitalization within 30 days before administration of the investigational product by discretion of the investigator.
5. Patients with a known clinically significant anemia (Hemoglobin <8.0 g/dL)
6. Patients with a known severe renal impairment (eGFR ≤ 30 mL/min/1.73 m2)
7. Patients with a known severe hepatic dysfunction
8. Patients with a known allergic reaction to the active ingredients (pyronaridine tetraphosphate, artesunate) and other ingredients of the investigational product
9. Patients with a gastrointestinal disease or who underwent a surgery that can affect the absorption, distribution, metabolism and excretion of the drug, or who have active gastritis, gastrointestinal tract/rectal bleeding, gastric ulcer, and pancreatitis or pancreatic function abnormalities (excluding general appendectomy or hernia repair surgery)
10. Patients who cannot be orally administered with the Investigational Product
11. Pregnant, breast-feeding or females with positive pregnancy test at screening
12. Females and males who have child-bearing plan or who are unwilling to commit to the use of the following methods of contraception* during study period and for 3 months after the study period
13. Patients who have participated in another clinical study/device study and received the investigational product/device within 28 days from signing the informed consent
14. Patients with Co-morbidity requiring surgery within 7 days before administration of the investigational product, or life-threatening co-morbidity within 30 days before administration of the investigational product
15. Patients with history of alcohol or drug abuse within 12 months before administration of the investigational product
16. Patients whom the investigator considers inappropriate for the study due to chronic underlying disease or other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1807 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects who require hospitalization or have died due to COVID-19 infection until post-dose D29. | follow up to Day29

SECONDARY OUTCOMES:
Time to sustained recovery (discharge) in hospitalized subjects (days) | follow up to Day29
29-day mortality after the first dose of the investigational product | Day29
11-point WHO clinical progression scale for clinical symptoms at D3, D7, D14, D21, and D29 after administration of the IP and changes compared to baseline | Day3, Day7, Day14, Day21, Day29
NEWS at D3, D7, D14, D21, and D29 after administration of the IP and changes compared to baseline | Day3, Day7, Day14, Day21, Day29
Percentage of subjects requiring acute therapy for more than 24 hours in a hospital or acute treatment facility or who have died due to COVID-19 until D29 after administration | follow up to Day29
Percentage of subjects who have newly diagnosed with pneumonia or aggravated pneumonia* according to baseline pneumonia criteria until D29 after administration of the IP | follow up to Day29
Change from baseline in COVID-19 viral load at D2, D3, D5, D7, and D14 | Day2, Day3, Day5, Day7, Day14
Percentage of subjects in the high-risk group** who require hospitalization or have died due to COVID-19 until post-dose D29 | follow up to Day29

CONTACTS AND LOCATIONS:
Locations (66):
- Argentina (6):
  - Instituto Medico Platense, Buenos Aires
  - Ciprec - Centro de Investigación Y Prevención Cardiovascular, Caba
  - Hospital de Agudos "Dr. Ignacio Pirovano", Caba
  - Instituto Médico Río Cuarto, Córdoba
  - Clinica Privada Independencia, Munro
  - Centro Médico IPAM, Santa Fe
- Chile (5):
  - Icegclinic, La Florida, Santiago Metropolitan
  - Clínica Universidad de los Andes, Las Condes, Santiago Metropolitan
  - Hospital Regional Dr. Leonardo Guzman de Antofagasta, Antofagasta
  - Centro de Estudios Clínicos e Investigaciones Médicas - CECIM, Santiago
  - IntegraMédica Las Condes, Santiago
- Colombia (13):
  - Clínica de la Costa Ltda, Barranquilla
  - Corazon IPS S.A.S, Barranquilla
  - IPS Centro Cientifico Asisitencial S.A.S, Barranquilla
  - Centro de Estudios e Investigación en salud-CEIS, Bogotá
  - Centro de Investigacion en Reumatología y Especialidades Médicas-CIREEM S.A.S, Bogotá
  - Fundación Valle del Lili, Cali
  - Institución Prestadora de servicios de salud Centro Medico Julian Coronel S.A.S, Cali
  - Clinica Universidad de la Sabana, Chía
  - Fundación Cardiovascular de Colombia, Floridablanca
  - Asociación IPS Médicos Internistas de Caldas S.A.S, Manizales
  - Healthy Medical Center S.A.S., Manizales
  - Programa de Estudio y Control de Enfermedades Tropicales PECET. Universidad de Antoquia, Medellín
  - Clinisalud del Sur S.A.S, Sabaneta
- Poland (7):
  - Krakowskie Centrum Medyczne, Krakow
  - Centrum Medyczne AMED Oddział w Łodzi, Lodz
  - NZOZ Le Med, Lodz
  - MEDICOME - Oświęcimskie Centrum Medyczne, Oświęcim
  - Przychodnia Lekarska Eskulap, Skierniewice
  - FutureMeds Warszawa Centrum, Warsaw
  - CMS Sp. z o.o., Wysokie Mazowieckie
- South Korea (33):
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si
  - Busan Medical Center, Busan
  - Keimyung University Dongsan Medical Center, Daegu
  - KyungPook National University Chilgok Hospital, Daegu
  - Kyungpook National University Hospital, Daegu
  - Chungnam national University Hospital, Daejeon
  - Chungnam National University Sejong Hospital, Daejeon
  - Gimpo Woori Hospital, Gimpo-si
  - Myongji Hospital, Goyang-si
  - Chonnam National University Bitgoeul Hospital, Gwangju
  - Gyeonggi Medical Center An-sung Hospital, Gyeonggi-do
  - Gyeonggi Medical Center Icheon Hospital, Gyeonggi-do
  - Gyeonggi Medical Center Paju Hospital, Gyeonggi-do
  - Gyeonggi Medical Center Pocheon Hospital, Gyeonggi-do
  - Gyeonggi Medical Center Suwon Hospital, Gyeonggi-do
  - Gyeonggi Medical Center Uijeongbu Hospital, Gyeonggi-do
  - Inje University Ilsan Paik Hospital, Ilsan
  - Incheon Sejong Hospital, Incheon
  - Inha University Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Pusan National University Hospital, Pusan
  - Boramae Medical Center, Seoul
  - Chosun University Hospital, Seoul
  - Chung-Ang University Hospital, Seoul
  - Eunpyeong St. Marys' Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Kyung Hee University Medical Center, Seoul
  - National Medical Center, Seoul
  - Sahmyook medical Center, Seoul
  - Seoul Medical Center, Seoul
  - Seoul Red Cross Hospital, Seoul
  - Ajou University Hospital, Suwon
  - Yongin Severance Hospital, Yŏngin
- United Kingdom (2):
  - Bridle Road Clinic (Liverpool), Birkenhead
  - Soho Road Health Centre, Birmingham